CLINICAL TRIAL: NCT05490810
Title: Effects of Trunk Stabilization Versus Activation Exercises on Pain and Disability in Postpartum Lumbo-pelvic Pain
Acronym: LPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0517
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Pelvic Pain
Keywords: Lumbo-pelvic Pain; Postpartum; Stabilization Exercises; Trunk Activation Exercises
MeSH Terms: conditions — Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk stabilization (Experimental): Trunk stabilization exercises were given three times a week for two weeks.
  Interventions: Other: Trunk stabilization
- Activation exercises (Experimental): Activation exercises exercises performed twice for 5s, with 2 min rest between them for three times a week for two weeks.
  Interventions: Other: Activation exercises

INTERVENTIONS:
Other: Trunk stabilization — Trunk stabilization exercises with
  * Static back: A roll of towel was pressed against the back and the position was held for 10 secs and then released
  * Static gluteus: The gluts were pressed inside and hold for 10 secs and then released.
  * Abdominal bracing: Brace your abdomen by contracting your entire abdomen. From here Perform different exercises such as raising your arms and then raising your legs.
  * Pelvic bridging: In crook lying, engage your gluts and trunk lift your hips towards the ceiling. Hold the position for 10 secs and then release.
  * SLR with-hold at 30 and 45 degrees: Ask the supine patient to raise the leg up-to 45 degrees and hold for 10 secs. Then raise the leg up-to 30 degrees then hold for 10 secs.
  Arms: Trunk stabilization
Other: Activation exercises — Activation exercises with
  * Upper rectus abdominis (URA) and lower rectus abdominis (LRA): body supine with hips and knees flexed 90°, with feet locked. Participants flexed the trunk (i.e. crunch execution) against resistance at the level of the shoulders..
  * External oblique (EO) and internal oblique (IO): side-lying with the hip at the edge of the bench and feet locked by a second operator. Participants performed side-bend exercise against resistance at the level of the shoulder.
  * Lower erector spinae (LES) and upper erector spinae (UES): prone position with ASIS at the edge of the bench and feet locked by a second operator. Participants performed a back extension against resistance at the level of the shoulders.
  Arms: Activation exercises

SUMMARY:
To compare the Effects of trunk stabilization versus activation exercises on pain and disability in postpartum lumbo-pelvic pain.

DETAILED DESCRIPTION:
Effects of stabilizing exercises on postpartum pelvic floor muscle function, lumbo-pelvic pain and disability. In results, stability exercises can help women with LPP enhance the function of their PFMs. Pregnancy and childbirth weakens PFMs and disrupts the load-transfer system in the lumbo-pelvic area. The use of PFMs in the right pattern can help these muscles operate better. Local stabilizing muscles are targeted during stabilization exercises, which increase pelvic motor control and stability.

As per researcher knowledge there was limited evidence present on the comparison of trunk stabilization and trunk activation exercises. Therefore, this study was conducted to find the effectiveness of trunk stabilization versus activation exercises on disability and pain in postpartum women with lumbo-pelvic pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* Female after postpartum
* Two or more positive posterior provocation test
* Active straight leg raises
* Pain onset during pregnancy

Exclusion Criteria:

* Orthopedic or rheumatologic disorders
* Intervertebral disc pathology
* Neoplasm or previuos surgery of spine
* History of fracture.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 2 weeks
  Pain intensity was assessed using a visual analog scale (VAS), which is a 100-mm ungraded line with two anchors. Its left and right anchors represented the minimum and maximum intensities of pain, respectively. The participants were asked to report their current pain intensity on the VAS.

SECONDARY OUTCOMES:
Oswestry disability index | 2 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools.

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam Muneeb, MS, Principal Investigator — Riphah International University
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaudhry RY, Muneeb HN, Amjad A, Shafique S, Naseem A, Shahzadi N. Comparing the effects of trunk stabilisation and activation exercises on pain and disability in postpartum lumbo-pelvic pain: A randomised controlled trial. J Pak Med Assoc. 2024 Jan;74(1):126-128. doi: 10.47391/JPMA.8395. PMID 38219179